CLINICAL TRIAL: NCT06491095
Title: A Randomized, Controlled, Cross-over Trial Examining the Effect of Flaxseed on Blood Cyanide Levels in Healthy Adults
Brief Title: Effect of Flax in Yogurt on Blood Cyanide Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Principal Investigator, Dr. Heather Blewett, Principle Investigator, St. Boniface Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 4030/4687
Record Dates: First submitted 2024-06-05; First posted 2024-07-08 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Flax; Blood Cyanide
MeSH Terms: interventions — Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- No Flax Product (Other): 175 g yogurt containing no flax product
  Interventions: Dietary Supplement: 0 g Flax
- 40 g whole ground flaxseed (Experimental): 175 g yogurt with 40 g whole ground flaxseed
  Interventions: Dietary Supplement: 40 g whole ground flaxseed
- 40 g roasted then ground whole flaxseed (Experimental): 175 g yogurt with 40 g roasted then ground whole flaxseed
  Interventions: Dietary Supplement: 40 g roasted then ground whole flaxseed
- 40 g of whole intact flaxseeds (Experimental): 175 g yogurt with 40 g of whole intact flaxseeds
  Interventions: Dietary Supplement: 40 g of whole intact flaxseeds
- 28 g flax hulls (Experimental): 175 g yogurt with 28 g flax hulls
  Interventions: Dietary Supplement: 28 g flax hulls

INTERVENTIONS:
Dietary Supplement: 0 g Flax — 175 g yogurt with no flax product
  Arms: No Flax Product
Dietary Supplement: 40 g whole ground flaxseed — 175 g yogurt with 40 g whole ground flaxseed
  Arms: 40 g whole ground flaxseed
Dietary Supplement: 40 g roasted then ground whole flaxseed — 175 g yogurt with 40 g roasted then ground whole flaxseed
  Arms: 40 g roasted then ground whole flaxseed
Dietary Supplement: 40 g of whole intact flaxseeds — 175 g yogurt with 40 g of whole intact flaxseeds
  Arms: 40 g of whole intact flaxseeds
Dietary Supplement: 28 g flax hulls — 175 g yogurt with 28 g flax hulls
  Arms: 28 g flax hulls

SUMMARY:
A randomized, controlled, cross-over post-prandial trial in healthy human volunteers will be conducted at the IH Asper Institute to determine the effect whole ground flaxseed, roasted then ground whole flaxseed, whole intact flaxseed and flaxseed hulls mixed into yogurt on blood cyanide levels.

DETAILED DESCRIPTION:
Participants will receive yogurt containing the following flaxseed products in a random order:

1. 40 g ground flaxseed, untreated;
2. 40 g ground flaxseed, roasted before grinding;
3. 40 g intact whole flaxseed;
4. 28 g flaxseed hulls;
5. 0 g flaxseed.

Venous blood will be collected at the following time points: 0 (before consumption of test product), 15, 30, 45, 60, 75, 90, 120, 150, 180 min.

Urine will be collected prior to consumption of test product and 180 min.

Primary endpoints: 1) Peak blood level of cyanide and incremental area under the curve (iAUC) for cyanide in blood over a 3h postprandial period. Secondary endpoint: 1) cyanogenic glycoside and thiocyanate concentrations in plasma and urine over a 3h postprandial period.

Tertiary endpoints: 1) metabolic profile in plasma and urine over 3 h postprandial period.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy adult, 18 years or older;
2. Willing to provide informed consent;
3. Willing/able to comply with the requirements of the study.

Exclusion Criteria:

1. Pregnant or lactating;
2. Medical history of disease that is currently under treatment;
3. Active treatment for any type of cancer within 1 year prior to study start;
4. Presence of a gastrointestinal disorder, daily use of any stomach acid-lowering medications or laxatives (including fibre supplements) within the past month or antibiotic use within the past 6 weeks;
5. Plasma concentration of vitamin B12 < 148 pmol/L;
6. Complete blood count outside normal range;
7. Medical history of liver disease or liver dysfunction (defined as plasma AST or ALT ≥3 times the upper limit of normal (ULN));
8. Fasting blood glucose ≥6.1 mmol/L and/or HbA1c ≥6.0%;
9. Fasting plasma total cholesterol >7.8 mmol/L;
10. Fasting plasma HDL <0.9 mmol/L;
11. Fasting plasma LDL >5.0 mmol/L;
12. Fasting plasma triglycerides >2.3 mmol/L;
13. Systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg;
14. Major surgery within the last 3 months;
15. Smoking, use of tobacco, vape or cannabis (within the last week);
16. Allergies to flaxseed or yogurt;
17. Aversion or unwillingness to eat study foods;
18. Participation in another clinical trial, current or in the past 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-16 (Estimated); Primary Completion 2025-03-28 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Peak blood level of cyanide | 180 minutes
  highest concentration of cyanide during 180 min postprandial period
iAUC blood cyanide | 180 min
  incremental area under the curve for cyanide from 0-180 min

SECONDARY OUTCOMES:
Cyanogenic glycoside and thiocyanate concentrations in plasma and urine | 180 minutes

OTHER OUTCOMES:
Concentration of metabolites in blood and urine | 180 minutes
  Identification and concentration of metabolites in plasma and urine determined by LC-QTOF-MS

CONTACTS AND LOCATIONS:
Overall Officials: Heather Blewett, PhD, Principal Investigator — Agriculture and Agri-Food Canada
Locations (1):
- I. H. Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Abraham K, Buhrke T, Lampen A. Bioavailability of cyanide after consumption of a single meal of foods containing high levels of cyanogenic glycosides: a crossover study in humans. Arch Toxicol. 2016 Mar;90(3):559-74. doi: 10.1007/s00204-015-1479-8. Epub 2015 Feb 24. PMID 25708890
- [Background] Agbor-Egbe T, Lape Mbome I. The effects of processing techniques in reducing cyanogen levels during the production of some Cameroonian cassava foods. Journal of Food Composition and Analysis. 2006 Jun;19(4):354-63.
- [Background] Carlsson L, Mlingi N, Juma A, Ronquist G, Rosling H. Metabolic fates in humans of linamarin in cassava flour ingested as stiff porridge. Food Chem Toxicol. 1999 Apr;37(4):307-12. doi: 10.1016/s0278-6915(99)00015-0. PMID 10418947
- [Background] Cressey P, Reeve J. Metabolism of cyanogenic glycosides: A review. Food Chem Toxicol. 2019 Mar;125:225-232. doi: 10.1016/j.fct.2019.01.002. Epub 2019 Jan 4. PMID 30615957
- [Background] Cressey P, Saunders D, Aupaau F. Evaluation of food safety risks associated with foods containing cyanogenic glycosides. New Zealand Food Safety Technical Paper No: 2022/29. 2022 Nov.
- [Background] Diaz-Rueda P, Morales de Los Rios L, Romero LC, Garcia I. Old poisons, new signaling molecules: the case of hydrogen cyanide. J Exp Bot. 2023 Oct 13;74(19):6040-6051. doi: 10.1093/jxb/erad317. PMID 37586035
- [Background] EFSA Panel on Contaminants in the Food Chain (CONTAM); Schrenk D, Bignami M, Bodin L, Chipman JK, Del Mazo J, Grasl-Kraupp B, Hogstrand C, Hoogenboom LR, Leblanc JC, Nebbia CS, Nielsen E, Ntzani E, Petersen A, Sand S, Vleminckx C, Wallace H, Benford D, Brimer L, Mancini FR, Metzler M, Viviani B, Altieri A, Arcella D, Steinkellner H, Schwerdtle T. Evaluation of the health risks related to the presence of cyanogenic glycosides in foods other than raw apricot kernels. EFSA J. 2019 Apr 11;17(4):e05662. doi: 10.2903/j.efsa.2019.5662. eCollection 2019 Apr. PMID 32626287
- [Background] Gleadow RM, Moller BL. Cyanogenic glycosides: synthesis, physiology, and phenotypic plasticity. Annu Rev Plant Biol. 2014;65:155-85. doi: 10.1146/annurev-arplant-050213-040027. Epub 2014 Feb 24. PMID 24579992
- [Background] Joint FAO/WHO Expert Committee on Food Additives (JECFA). Safety evaluation of certain food additives and contaminants. WHO food additives series; 65. 2012
- [Background] Mazza G and Oomah BD. Flaxseed, dietary fiber, and cyanogens. In: "Flaxseed in human nutrition", Editors: Cunnane, S.C. and Thompson, L.U., AOCS Press, 1995 56-81.
- [Background] Muir AD, Westcott ND. Quantitation of the lignan secoisolariciresinol diglucoside in baked goods containing flax seed or flax meal. J Agric Food Chem. 2000 Sep;48(9):4048-52. doi: 10.1021/jf990922p. PMID 10995312
- [Background] Ngudi DD, Kuo YH, Lambein F. Cassava cyanogens and free amino acids in raw and cooked leaves. Food Chem Toxicol. 2003 Aug;41(8):1193-7. doi: 10.1016/s0278-6915(03)00111-x. PMID 12842188
- [Background] Parikh M, Netticadan T, Pierce GN. Flaxseed: its bioactive components and their cardiovascular benefits. Am J Physiol Heart Circ Physiol. 2018 Feb 1;314(2):H146-H159. doi: 10.1152/ajpheart.00400.2017. Epub 2017 Nov 3. PMID 29101172
- [Background] Yulvianti M, Zidorn C. Chemical Diversity of Plant Cyanogenic Glycosides: An Overview of Reported Natural Products. Molecules. 2021 Jan 30;26(3):719. doi: 10.3390/molecules26030719. PMID 33573160
- See also: New Zealand Food Safety Authority. Cyanogenic glycosides -Information sheet. — https://www.mpi.govt.nz/dmsdocument/25688/direct
- See also: Schneider B. Activity of β-glucosidase in plants with high content of cyanogenic glycosides as important factor determining their toxicity. Toxicology Letters. 2014 229, S170-S170 — https://doi.org/10.1016/j.toxlet.2014.06.582